CLINICAL TRIAL: NCT01363388
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of CCX168 in Subjects With Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis on Background of Cyclophosphamide or Rituximab Treatment
Brief Title: A Study to Evaluate the Safety and Efficacy of CCX168 in Subjects With ANCA-Associated Vasculitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL002_168
Record Dates: First submitted 2011-05-26; First posted 2011-06-01 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Vasculitis
MeSH Terms: conditions — Vasculitis | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo plus a full dose of oral glucocorticoids for steps 1 and 2 of the study
  Interventions: Drug: Placebo
- CCX168 (Experimental): 30 mg Active study medication, plus either two-thirds reduced dose of oral glucocorticoids for step 1 of the study, or no oral glucocorticoids for step 2 of the study
  Interventions: Drug: CCX168

INTERVENTIONS:
Drug: Placebo — BID for 84 days
  Arms: Placebo
Drug: CCX168 — BID for 84 days
  Arms: CCX168

SUMMARY:
The aim of this trial is to optimize the treatment to induce remission for patients with non-life-threatening anti-neutrophil cytoplasmic antibody vasculitis (AAV). The intent is to reduce the toxicity of induction therapy by reducing the overall exposure to or eliminating entirely the use of systemic corticosteroids during the induction period with an inhibitor of the complement C5a receptor plus cyclophosphamide or rituximab.

DETAILED DESCRIPTION:
The primary safety objective of this study is to evaluate the safety and tolerability of CCX168 in subjects with AAV on background cyclophosphamide or rituximab treatment.

The primary efficacy objective is to evaluate the efficacy of CCX168 based on the Birmingham Vasculitis Activity Score (BVAS) version 3.

The secondary objectives of this study include assessment of the feasibility of reducing or eliminating the use of corticosteroids in the treatment of subjects with ANCA-associated vasculitis without the need for rescue corticosteroid measures and the effect of CCX168 on several disease parameters.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis or renal limited vasculitis
* Male and postmenopausal or surgically sterile female subjects aged at least 18 years with new or relapsed AAV where treatment with cyclophosphamide or rituximab would be required
* Positive indirect immunofluorescence (IIF) test for P-ANCA or C-ANCA, or positive ELISA test for anti-proteinase-3 (PR3) or anti-myeloperoxidase (MPO) at screening
* Estimated glomerular filtration rate (eGFR) ≥ 20mL/min
* Have at least one "major" item, or at least 3 non-major items, or at least 2 renal items on the BVAS version 3

Key Exclusion Criteria:

* Severe disease as determined by rapidly progressive glomerulonephritis, alveolar hemorrhage, hemoptysis, rapid-onset mononeuritis multiplex or central nervous system involvement
* Any other multi-system autoimmune disease
* Medical history of coagulopathy or bleeding disorder
* Received cyclophosphamide within 12 weeks of screening; if on azathioprine, mycophenolate mofetil or methotrexate at the time of screening, these drugs must be withdrawn prior to receiving the cyclophosphamide or rituximab dose on Day 1
* Received high-dose intravenous corticosteroids within 4 weeks of screening
* On an oral dose of a corticosteroid of more than 10mg prednisone-equivalent at the time of screening
* Received rituximab or other B-cell antibody within 52 weeks of screening or 26 weeks provided B cell reconstitution has occurred; received anti-TNF treatment, abatacept, alemtuzumab, IVIg or plasma exchange within 12 weeks of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- Austria (3):
  - Feldkirch
  - Innsbruck
  - Linz
- Belgium (6):
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Prague, Czechia
- France (9):
  - Bordeaux
  - Boulogne-sur-Mer
  - Brest
  - Colmar
  - Grenoble
  - Nantes
  - Paris
  - Saint-Jacques
  - Valenciennes
- Germany (6):
  - Berlin
  - Cologne
  - Dresden
  - Freiburg im Breisgau
  - Fulda
  - Heidelberg
- Budapest, Hungary
- Netherlands (4):
  - Groningen
  - Leiden
  - Rotterdam
  - Utrecht
- Poland (4):
  - Bialystok
  - Katowice
  - Szczecin
  - Wroclaw
- Sweden (4):
  - Linköping
  - Lund
  - Malmo
  - Stockholm
- United Kingdom (6):
  - Birmingham
  - Cambridge
  - London
  - Manchester
  - Oxford
  - Reading

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Cravedi P, Leventhal J, Lakhani P, Ward SC, Donovan MJ, Heeger PS. Immune cell-derived C3a and C5a costimulate human T cell alloimmunity. Am J Transplant. 2013 Oct;13(10):2530-9. doi: 10.1111/ajt.12405. Epub 2013 Sep 6. PMID 24033923
- See also: Randomized Trial of C5a Receptor Inhibitor Avacopan in ANCA-Associated Vasculitis — https://jasn.asnjournals.org/content/28/9/2756

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo BID Plus 60 mg Prednisone: Drug: Placebo BID plus 60 mg prednisone
- CCX168 30 mg BID Plus 20 mg Prednisone: Drug: CCX168 30 mg BID plus 20 mg prednisone
- CCX168 30 mg BID Without Prednisone: Drug: CCX168 30 mg BID without prednisone
Period: Overall Study
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Started | 23 | 22 | 22
Completed | 18 | 19 | 18
Not Completed | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone | Total
Number analyzed (Participants) | 23 | 22 | 22 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (14.0) | 57.0 (14.2) | 57.4 (14.0) | 57.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 6 | 20
  Male | 17 | 14 | 16 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 22 | 22 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 23 | 22 | 22 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 3 | 2 | 4 | 9
  Past Smoker | 11 | 6 | 8 | 25
  Never Smoked | 9 | 14 | 10 | 33
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index Population: Values provided for subjects with measurements at baseline
  kg/m^2
    number analyzed (Participants) | 23 | 21 | 21 | 65
    (all) | 27.3 (7.09) | 24.9 (4.05) | 26.5 (4.66) | 26.3 (5.49)
ANCA disease status [Count of Participants; unit: Participants] — ANCA = anti-neutrophil cytoplasmic antibody
  Participants
    Newly diagnosed | 18 | 15 | 16 | 49
    Relapsed | 5 | 7 | 6 | 18
ANCA- associated vasculitis disease duration at screening [Median (Full Range); unit: months] — ANCA = anti-neutrophil cytoplasmic antibody Population: Values provided for subjects with measurements at baseline
  months
    number analyzed (Participants) | 23 | 22 | 21 | 66
    (all) | 0.0 [0 to 162] | 0.0 [0 to 61] | 1.0 [0 to 108] | 0.0 [0 to 162]
Background treatment [Count of Participants; unit: Participants]
  Rituximab | 3 | 5 | 5 | 13
  Cyclophosphamide | 20 | 17 | 17 | 54
Type of AAV [Count of Participants; unit: Participants] — AAV= ANCA-associated vasculitis GPA = granulomatosis with polyangitis (Wegener's)
  Participants
    GPA | 10 | 11 | 12 | 33
    Microscopic polyangiitis | 10 | 9 | 9 | 28
    Renal-limited vasculitis | 2 | 2 | 1 | 5
    Unknown | 1 | 0 | 0 | 1
ANCA status categorical [Count of Participants; unit: Participants] — ANCA = anti-neutrophil cytoplasmic antibody MPO=myeloperoxidase PR3=proteinase 3
  Participants
    Anti-MPO positive | 10 | 12 | 13 | 35
    Anti-PR3 positive | 11 | 10 | 8 | 29
    Both anti-MPO positive and anti-PR3 positive | 1 | 0 | 0 | 1
    ANCA equivocal | 0 | 0 | 1 | 1
    ANCA negative | 1 | 0 | 0 | 1
BVAS total score [Mean (Standard Deviation); unit: units on a scale] — The Birmingham Vasculitis Activity Score (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
  units on a scale | 13.2 (5.80) | 14.3 (5.98) | 13.8 (6.38) | 13.7 (5.98)
VDI score [Mean (Standard Deviation); unit: units on a scale] — The Vasculitis Damage Index (VDI) is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health)
  units on a scale | 1.2 (1.35) | 0.9 (1.46) | 0.5 (1.19) | 0.9 (1.35)
Glomerular filtration rate (MDRD) [Mean (Standard Deviation); unit: mL/min/1.73 m2] — MDRD=Modification of Diet in Renal Disease Population: Values provided for subjects with measurements at baseline
  mL/min/1.73 m2
    number analyzed (Participants) | 22 | 22 | 22 | 66
    (all) | 47.6 (15.08) | 52.5 (26.70) | 54.7 (19.64) | 51.6 (20.92)
Albumin: creatinine ratio [Geometric Mean (Full Range); unit: mg/g] — Population: Values provided for subjects with measurements at baseline
  mg/g
    number analyzed (Participants) | 22 | 22 | 21 | 65
    (all) | 353.9 [28 to 5962] | 278.6 [24 to 2459] | 283.4 [25 to 3051] | 303.8 [24 to 5962]
Urinary MCP-1 : creatinine ratio [Geometric Mean (Full Range); unit: pg/mg creatinine] — MCP-1 = Monocyte chemoattractant protein 1
  pg/mg creatinine | 825.9 [171.2 to 2549.2] | 1266.1 [360.8 to 7290.5] | 846.4 [107.2 to 6075.7] | 957.9 [107.2 to 7290.5]
Urinary red blood cells [Count of Participants; unit: Participants] — HPF= high power field
  Participants
    30-49 per hpf | 6 | 4 | 2 | 12
    50-75 per hpf | 5 | 4 | 3 | 12
    >75 per hpf | 3 | 5 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Disease Response at Day 85
Description: Disease response is defined as BVAS percentage reduction from baseline of at least 50% plus no worsening in any body system component.
Time Frame: Baseline to Day 85
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 22 | 21
proportion of participants | 0.7 | 0.86 | 0.81

2. Secondary Outcome: Proportion of Patients Achieving Renal Response at Day 85
Description: Renal response, assessed in patients with hematuria and albuminuria at baseline, and defined as an improvement in renal parameters, i.e., an increase from baseline to Day 85 in eGFR (Estimated glomerular filtration rate), MDRD (Modification of Diet in Renal Disease), serum creatinine equation, a decrease from baseline to Day 85 in haematuria (central laboratory microscopic count of urinary red blood cells) , decrease from baseline to Day 85 in albuminuria count (first morning UACR (urinary albumin:creatinine ratio).
Time Frame: Baseline to Day 85
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 18 | 18
proportion of participants | 0.4 | 0.56 | 0.33

3. Secondary Outcome: Proportion of Subjects Achieving Disease Remission at Day 85
Description: Disease remission is defined as BVAS (Birmingham Vasculitis Activity Score) of 0 or 1 plus no worsening in eGFR (Estimated glomerular filtration rate) and urinary RBC (Red Blood cell) count <10/high power field (hpf)
Time Frame: Day 85
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 22 | 21
proportion of participants | 0.35 | 0.27 | 0.19

4. Secondary Outcome: Percent Change From Baseline to Day 85 in BVAS
Description: Percent change in Burmingham Vasculitis Index Score (BVAS) at week 12, higher percentage change indicates worse outcome
  BVAS = Birmingham Vasculitis Activity Score
  The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health). A negative percentage change indicated improvement in health.
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 19 | 20 | 19
percentage change | -56.45 (62.100) | -79.05 (23.005) | -73.01 (29.464)

5. Secondary Outcome: Change From Baseline to Day 85 in eGFR
Description: eGFR (Estimated glomerular filtration rate) based on the MDRD (Modification of Diet in Renal Disease) formula using serum creatinine
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 21 | 19
ml/min/1.73 m^2 | 5.55 (10.211) | 6.00 (10.469) | 0.79 (9.549)

6. Secondary Outcome: Percent Change From Baseline to Day 85 in eGFR
Description: as for outcome 5
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 21 | 19
percentage change | 15.36 (23.685) | 19.91 (23.034) | 0.92 (20.562)

7. Secondary Outcome: Proportion of Subjects Achieving Urinary RBC Count <=5/Hpf at Any Time During the 84-day Treatment Period
Description: In subjects with baseline hematuria >5 RBCs/hpf (Red Blood Cell/High Power Field)
Time Frame: Baseline to Day 85
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 19 | 18 | 18
proportion of participants | 0.79 | 0.61 | 0.61

8. Secondary Outcome: Time to First Achieving Urinary RBC Count <=5/Hpf at Any Point During the 84-day Treatment Period
Description: In subjects with baseline hematuria <=5 RBCs/hpf (Red Blood Cell/High Power Field)
Time Frame: Baseline to Day 85
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 19 | 18 | 18
days | 69.0 [28.0 to 84.0] | 69.0 [27.0 to NA] — Insufficient number of participants with events to estimate 75th quantile | 42.0 [7.0 to NA] — Insufficient number of participants with events to estimate 75th quantile

9. Secondary Outcome: Proportion of Subjects Achieving Urinary RBC Count <30/Hpf at Any Time During the 84-day Treatment Period
Description: In subjects with baseline hematuria >=30 RBCs/hpf,(Red Blood Cell/High Power Field)
Time Frame: Baseline to Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 12 | 13 | 7
Participants | 11 | 13 | 5

10. Secondary Outcome: Time to First Achieving Urinary RBC Count <=30/Hpf at Any Point During the 84-day Treatment Period
Description: In subjects with baseline hematuria <=30 RBCs/hpf (Red Blood Cell/High Power Field)
Time Frame: Baseline to Day 85
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 11 | 13 | 7
days | 10.5 [1.0 to 35.0] | 21.0 [7.0 to 42.0] | 42.0 [1.0 to NA] — Insufficient number of participants with events to estimate 75th quantile

11. Secondary Outcome: Percent Change From Baseline to Day 85 in Urinary RBC Count
Description: In subjects with hematuria at baseline, RBC (Red Blood Cell)
Time Frame: Baseline to day 85
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 19 | 17
percentage change | -72.37 [-99.4 to 66.7] | 1.63 [-99.7 to 1150.0] | -21.26 [-99.4 to 368.8]

12. Secondary Outcome: Percent Change From Baseline to Day 85 in UACR
Description: In subjects with albuminuria at baseline UACR (urinary albumin:creatinine ratio)
Time Frame: Baseline to Day 85
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 20 | 18
percentage change | -3.10 [-71.1 to 131.7] | -34.18 [-89.2 to 173.1] | -15.21 [-85.9 to 360.3]

13. Secondary Outcome: Percent Change From Baseline to Day 85 in Urinary MCP-1:Creatinine Ratio
Description: Urinary Monocyte Chemoattractant Protein-1 (MCP-1):creatinine ratio
Time Frame: Baseline to Day 85
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 20 | 19
percentage change | -37.57 [-72.7 to 41.0] | -59.29 [-93.6 to 60.1] | -39.44 [-90.7 to 59.0]

14. Secondary Outcome: Proportion of Subjects Requiring Rescue IV or Oral Glucocorticoid Treatment
Time Frame: Baseline to Day 85
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 11 | 9 | 8
proportion of participants | 0 | 0.33 | 0.13

15. Secondary Outcome: Change From Baseline to Day 85 in the Vasculitis Damage Index
Description: VDI=Vasculitis Damage Index; The VDI is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health).
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 0.7 (0.81) | 0.3 (0.57) | 0.2 (0.54)

16. Secondary Outcome: Change From Baseline to Day 85 in Health-related Quality of Life as Measured by the SF-36 v2
Description: SF-36v2: Medical Outcomes Survey Short Form-36 version 2. SF-36v2 measures each of the following eight health domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Scores on each item are summed and averaged. The SF-36v2 component domain scores range from 0 (worst health) to 100 (best health).
Time Frame: Baseline, Day 29 & Day 85
Population: Number of subjects with data at baseline and the specified visit are specified.
Measure: Mean (Standard Error); unit: Change from baseline score on a scale
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 10 | 14 | 8
Change from baseline score on a scale
  SF-36 Role Physical (Day 29): number analyzed (Participants) | 9 | 14 | 8
  SF-36 Role Physical (Day 29) | 9.7 (10.73) | 13.8 (7.61) | 8.6 (6.02)
  SF-36 Role Physical (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Role Physical (Day 85) | 13.7 (11.06) | 36.1 (9.28) | 16.1 (9.24)
  SF-36 Bodily pain (Day 29): number analyzed (Participants) | 9 | 13 | 8
  SF-36 Bodily pain (Day 29) | 3.1 (10.63) | 17.3 (8.42) | 5.1 (16.75)
  SF-36 Bodily pain (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Bodily pain (Day 85) | 12.8 (7.36) | 21.7 (9.54) | 14.0 (9.30)
  SF-36 General Health Perceptions (Day 29): number analyzed (Participants) | 9 | 13 | 8
  SF-36 General Health Perceptions (Day 29) | 2.5 (8.26) | 3.7 (4.60) | -13.7 (10.21)
  SF-36 General Health Perceptions (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 General Health Perceptions (Day 85) | 5.7 (6.05) | 2.3 (3.93) | -1.5 (5.51)
  SF-36 Vitality (Day 29): number analyzed (Participants) | 9 | 13 | 8
  SF-36 Vitality (Day 29) | 7.63 (6.403) | 12.98 (7.400) | -0.78 (3.630)
  SF-36 Vitality (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Vitality (Day 85) | 4.36 (6.457) | 22.28 (7.541) | 10.71 (5.893)
  SF-36 Social Functioning (Day 29): number analyzed (Participants) | 9 | 14 | 8
  SF-36 Social Functioning (Day 29) | -2.8 (11.74) | 24.1 (6.07) | -7.8 (6.22)
  SF-36 Social Functioning (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Social Functioning (Day 85) | 6.3 (9.90) | 35.6 (6.91) | 5.4 (3.72)
  SF-36 Mental Health (Day 29): number analyzed (Participants) | 9 | 13 | 8
  SF-36 Mental Health (Day 29) | 1.7 (2.20) | 10.8 (3.71) | -8.1 (6.88)
  SF-36 Mental Health (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Mental Health (Day 85) | -1.0 (4.88) | 16.5 (4.65) | 2.1 (4.86)
  SF-36 Reported Health Transition (Day 29): number analyzed (Participants) | 9 | 14 | 8
  SF-36 Reported Health Transition (Day 29) | 0.2 (0.22) | -0.6 (0.41) | 0.3 (0.31)
  SF-36 Reported Health Transition (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Reported Health Transition (Day 85) | 0.0 (0.37) | -1.2 (0.48) | -0.4 (0.48)
  SF-36 Physical Functioning (Day 29): number analyzed (Participants) | 9 | 14 | 8
  SF-36 Physical Functioning (Day 29) | 5.0 (6.18) | 7.0 (6.90) | 8.2 (11.46)
  SF-36 Physical Functioning (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Physical Functioning (Day 85) | 5.2 (7.00) | 13.5 (7.73) | 11.4 (8.43)
  SF-36 Role-Emotional (Day 29): number analyzed (Participants) | 9 | 14 | 8
  SF-36 Role-Emotional (Day 29) | 1.9 (9.08) | 20.3 (8.04) | -1.1 (8.97)
  SF-36 Role-Emotional (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Role-Emotional (Day 85) | 0.0 (10.98) | 21.8 (9.42) | 10.7 (8.27)
  SF-36 Physical Component Summary (Day 29): number analyzed (Participants) | 9 | 12 | 8
  SF-36 Physical Component Summary (Day 29) | 2.693 (3.436) | 4.074 (2.601) | 2.826 (4.526)
  SF-36 Physical Component Summary (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Physical Component Summary (Day 85) | 5.383 (2.694) | 6.744 (3.132) | 4.863 (2.415)
  SF-36 Mental Health Summary (Day 29): number analyzed (Participants) | 9 | 12 | 8
  SF-36 Mental Health Summary (Day 29) | 0.303 (3.120) | 10.855 (3.244) | -4.760 (3.266)
  SF-36 Mental Health Summary (Day 85): number analyzed (Participants) | 10 | 13 | 7
  SF-36 Mental Health Summary (Day 85) | -0.766 (3.888) | 11.779 (3.428) | 2.197 (1.066)

17. Secondary Outcome: Change From Baseline to Day 85 in Health-related Quality of Life as Measured by the EQ-5D-5L
Description: EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given can be converted into an Index Score ranging from 0 for death to 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Baseline, Day 29 and Day 85
Population: Number of subjects with data at baseline and the specified visit are specified.
Measure: Mean (Standard Deviation); unit: Change from baseline score on a scale
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
Number analyzed (Participants) | 9 | 13 | 9
Change from baseline score on a scale
  VAS Score (Day 29): number analyzed (Participants) | 9 | 13 | 8
  VAS Score (Day 29) | -2.4 (10.61) | 6.5 (17.96) | 4.5 (12.62)
  VAS Score (Day 85): number analyzed (Participants) | 9 | 13 | 7
  VAS Score (Day 85) | -3.3 (13.23) | 11.8 (17.61) | 4.0 (4.69)
  Index Score (Day 29): number analyzed (Participants) | 9 | 13 | 8
  Index Score (Day 29) | -0.044 (0.1597) | 0.034 (0.1111) | -0.057 (0.0952)
  Index Score (Day 85): number analyzed (Participants) | 9 | 13 | 7
  Index Score (Day 85) | -0.043 (0.1718) | 0.067 (0.1314) | -0.047 (0.0721)

ADVERSE EVENTS:
Time Frame: 168 Day Treatment Period
Description: An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication
Arm/Group | Placebo BID Plus 60 mg Prednisone | CCX168 30 mg BID Plus 20 mg Prednisone | CCX168 30 mg BID Without Prednisone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/23 | 8/22 | 10/22
Other Adverse Events (participants affected / at risk) | 21/23 | 21/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID Plus 60 mg Prednisone (N=23) | CCX168 30 mg BID Plus 20 mg Prednisone (N=22) | CCX168 30 mg BID Without Prednisone (N=22)
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Febrile Infection (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2
Viral Infection (Infections and infestations) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1
Pancreatic Enzyme Increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal Impairement (Renal and urinary disorders) | 0 | 1 | 1
Renal Vasculitis (Renal and urinary disorders) | 1 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Microscopic Polyangiitis (Vascular disorders) | 0 | 0 | 1
Vasculitius (Vascular disorders) | 1 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID Plus 60 mg Prednisone (N=23) | CCX168 30 mg BID Plus 20 mg Prednisone (N=22) | CCX168 30 mg BID Without Prednisone (N=22)
Nasopharyngitis (Infections and infestations) | 5 | 4 | 5
Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 2
Rhinitis (Infections and infestations) | 1 | 2 | 2
Oral Herpes (Infections and infestations) | 1 | 0 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0
Viral Infection (Infections and infestations) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 7 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3
Constipation (Gastrointestinal disorders) | 5 | 3 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Muscle Spams (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 3
Fatigue (General disorders) | 3 | 0 | 4
Oedema Peripheral (General disorders) | 5 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 3 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 2
Breath Sounds Abnormal (Investigations) | 2 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 6
Vasculitis (Vascular disorders) | 2 | 3 | 2
Deep Vein Thrombosis (Vascular disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 4
Paraesthesia (Nervous system disorders) | 3 | 3 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 3 | 0
Renal Vasculitis (Renal and urinary disorders) | 2 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 1 | 1

LIMITATIONS AND CAVEATS:
This study is relatively small and the treatment duration was short.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-09-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT01363388/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT01363388/SAP_001.pdf